CLINICAL TRIAL: NCT03409276
Title: A Phase 1 Clinical Trial to Evaluate the Safety and Immunogenicity of Polyvalent Env (A,B,C,A/E) / Gag (C) DNA and gp120 (A,B,C,A/E) Protein/GLA-SE HIV-1 Vaccines (PDPHV-201401) as a Prime-boost Regimen or Co-administered in Repeated Doses, in Healthy, HIV-1-Uninfected Adult Participants
Brief Title: Evaluating the Safety and Immunogenicity of Env (A,B,C,A/E)/Gag (C) DNA and gp120 (A,B,C,A/E) Protein/GLA-SE HIV Vaccines, Given Individually or Co-administered, in Healthy, HIV-1-Uninfected Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HVTN 124; 38302 (Registry Identifier: DAIDS-ES Registry Number)
Record Dates: First submitted 2018-01-09; First posted 2018-01-24 (Actual); Results first posted 2022-04-25 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-03

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — Genes, env; Vaccines, DNA; Plasmids; HIV Envelope Protein gp120; glucopyranosyl lipid-A

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Group 1 (Treatment): Protein Vaccine/GLA-SE (Experimental): Participants will receive 400 mcg of gp120 (A,B,C,A/E) protein vaccine admixed with GLA-SE adjuvant at Day 0 and Month 2.
  Interventions: Biological: gp120 (A,B,C,A/E) Protein Vaccine; Biological: GLA-SE adjuvant
- Group 1 (Control) (Placebo Comparator): Participants will receive placebo at Day 0 and Month 2.
  Interventions: Biological: Placebo
- Group 2 (Treatment) DNA Vaccine+Placebo+Protein Vaccine/GLA-SE (Experimental): Participants will receive 2 mg of env (A,B,C,A/E)/gag (C) DNA vaccine and placebo at Day 0 and Months 1 and 3. Participants will receive 400 mcg of gp120 (A,B,C,A/E) protein vaccine admixed with GLA-SE adjuvant and a placebo vaccine at Months 6 and 8.
  Interventions: Biological: env (A,B,C,A/E)/gag (C) DNA Vaccine; Biological: gp120 (A,B,C,A/E) Protein Vaccine; Biological: Placebo; Biological: GLA-SE adjuvant
- Group 2 (Control) (Placebo Comparator): Participants will receive placebo at Day 0 and Months 1, 3, 6, and 8.
  Interventions: Biological: Placebo
- Group 3 (Treatment): DNA Vaccine+Protein Vaccine/GLA-SE (Experimental): Participants will receive 2 mg of the env (A,B,C,A/E)/gag (C) DNA vaccine and 400 mcg of gp120 (A,B,C,A/E) protein vaccine admixed with GLA-SE adjuvant at Day 0 and Months 1, 3, 6, and 8.
  Interventions: Biological: env (A,B,C,A/E)/gag (C) DNA Vaccine; Biological: gp120 (A,B,C,A/E) Protein Vaccine; Biological: GLA-SE adjuvant
- Group 3 (Control) (Placebo Comparator): Participants will receive placebo at Day 0 and Months 1, 3, 6, and 8.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: env (A,B,C,A/E)/gag (C) DNA Vaccine — Administered by intramuscular injection in the deltoid.
  Other Names: Polyvalent DNA (PDPHV-201401) Plasmid
  Arms: Group 2 (Treatment) DNA Vaccine+Placebo+Protein Vaccine/GLA-SE; Group 3 (Treatment): DNA Vaccine+Protein Vaccine/GLA-SE
Biological: gp120 (A,B,C,A/E) Protein Vaccine — Administered by intramuscular injection in the deltoid.
  Other Names: PDPHV-201401 Recombinant Proteins gp120A, gp120B, gp120C, gp120AE
  Arms: Group 1 (Treatment): Protein Vaccine/GLA-SE; Group 2 (Treatment) DNA Vaccine+Placebo+Protein Vaccine/GLA-SE; Group 3 (Treatment): DNA Vaccine+Protein Vaccine/GLA-SE
Biological: Placebo — Sodium Chloride for Injection, USP 0.9%; Administered by intramuscular injection in the deltoid.
  Arms: Group 1 (Control); Group 2 (Control); Group 2 (Treatment) DNA Vaccine+Placebo+Protein Vaccine/GLA-SE; Group 3 (Control)
Biological: GLA-SE adjuvant — Administered by intramuscular injection in the deltoid.
  Other Names: glucopyranosyl lipid adjuvant-stable emulsion
  Arms: Group 1 (Treatment): Protein Vaccine/GLA-SE; Group 2 (Treatment) DNA Vaccine+Placebo+Protein Vaccine/GLA-SE; Group 3 (Treatment): DNA Vaccine+Protein Vaccine/GLA-SE

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and immunogenicity of env (A,B,C,A/E)/gag (C) DNA and gp120 (A,B,C,A/E) protein/GLA-SE HIV-1 vaccines (PDPHV-201401) as a prime-boost regimen or co-administered in repeated doses, in healthy, HIV-1-uninfected adults.

DETAILED DESCRIPTION:
This study will evaluate the safety, tolerability, and immunogenicity of env (A,B,C,A/E)/gag (C) DNA and gp120 (A,B,C,A/E) protein/GLA-SE HIV-1 vaccines (PDPHV-201401) as a prime-boost regimen or co-administered in repeated doses, in healthy, HIV-1-uninfected adults.

The study will be conducted in two parts (Part A and Part B).

Participants in Part A will be randomly assigned to either Group 1 (Treatment) or Group 1 (Control). Participants in Group 1 (Treatment) will receive the gp120 (A,B,C,A/E) protein vaccine admixed with GLA-SE adjuvant on Day 0 and Month 2. Participants in Group 1 (Control) will receive placebo on Day 0 and Month 2.

Researchers will evaluate study data from Part A before enrolling participants in Part B.

Participants in Part B will be enrolled in either Groups 2 or 3. Within Group 2, participants will be randomly assigned to either Group 2 (Treatment) or Group 2 (Control). Participants in Group 2 (Treatment) will receive the env (A,B,C,A/E)/gag (C) DNA vaccine and placebo on Day 0 and Months 1 and 3. At Months 6 and 8, participants will receive the gp120 (A,B,C,A/E) protein vaccine admixed with GLA-SE adjuvant and a placebo vaccine. Participants in Group 2 (Control) will receive placebo on Day 0 and Months 1, 3, 6, and 8.

Participants in Group 3 will be randomly assigned to either Group 3 (Treatment) or Group 3 (Control). Participants in Group 3 (Treatment) will receive the env (A,B,C,A/E)/gag (C) DNA vaccine and the gp120 (A,B,C,A/E) protein vaccine admixed with GLA-SE adjuvant on Day 0 and Months 1, 3, 6, and 8. Participants in Group 3 (Control) will receive placebo on Day 0 and Months 1, 3, 6, and 8.

Study visits for participants in Part A will occur on Day 0, Week 2, and Months 2, 2.5, 5, and 8. Study visits for participants in Part B will occur on Day 0, Week 2, and Months 1, 1.5, 3, 3.5, 6, 6.5, 8, 8 + 1 Week, 8.5, 11, and 14. Visits may include physical examinations, blood and urine collection, HIV testing, risk reduction counseling, and questionnaires. Participants in Part B may also have optional saliva, semen, cervical fluid, rectal fluid, and stool sample collection.

Study staff will contact all participants 12 months after the last vaccination for follow-up health monitoring.

ELIGIBILITY:
Inclusion Criteria:

General and Demographic Criteria

* Age of 18 to 50 years
* Access to a participating HIV Vaccine Trials Network (HVTN) clinical research site (CRS) and willingness to be followed for the planned duration of the study
* Ability and willingness to provide informed consent
* Assessment of understanding: volunteer demonstrates understanding of this study; completes a questionnaire prior to first vaccination with verbal demonstration of understanding of all questionnaire items answered incorrectly
* Willing to be contacted 12 months after the last vaccination
* Agrees not to enroll in another study of an investigational research agent
* Good general health as shown by medical history, physical exam, and screening laboratory tests

HIV-Related Criteria:

* Willingness to receive HIV test results
* Willingness to discuss HIV infection risks and amenable to HIV risk reduction counseling.
* Assessed by the clinic staff as being at "low risk" for HIV infection and committed to maintaining behavior consistent with low risk of HIV exposure through the last required protocol clinic visit.

Laboratory Inclusion Values

Hemogram/Complete Blood Count (CBC)

* Hemoglobin greater than or equal to 11.0 g/dL for volunteers who were born female, greater than or equal to 13.0 g/dL for volunteers who were born male
* White blood cell count equal to 3,300 to 12,000 cells/mm^3
* Total lymphocyte count greater than or equal to 800 cells/mm^3
* Remaining differential either within institutional normal range or with site physician approval
* Platelets equal to 125,000/mm^3 to 450,000/mm^3

Chemistry

* Chemistry panel: Alanine aminotransferase (ALT), aspartate aminotransferase (AST), and alkaline phosphatase less than 1.25 times the institutional upper limit of normal; creatinine less than or equal to institutional upper limit of normal.

Virology

* Negative HIV-1 and -2 blood test: US volunteers must have a negative US Food and Drug Administration (FDA)-approved enzyme immunoassay (EIA).
* Negative Hepatitis B surface antigen (HBsAg)
* Negative anti-Hepatitis C virus antibodies (anti-HCV), or negative HCV polymerase chain reaction (PCR) if the anti-HCV is positive

Urine

* Normal urine:

  * Negative urine glucose, and
  * Negative or trace urine protein, and
  * Negative or trace urine hemoglobin (if trace hemoglobin is present on dipstick, a microscopic urinalysis with red blood cells levels within institutional normal range).

Reproductive Status

* Volunteers who were born female: negative serum or urine beta human chorionic gonadotropin (β-HCG) pregnancy test performed prior to vaccination on the day of initial vaccination. Persons who are NOT of reproductive potential due to having undergone total hysterectomy or bilateral oophorectomy (verified by medical records), are not required to undergo pregnancy testing.
* Reproductive status: A volunteer who was born female must:

  * Agree to consistently use effective contraception (see the protocol for more information) for sexual activity that could lead to pregnancy from at least 21 days prior to enrollment until after the last required protocol clinic visit. Effective contraception is defined as using the following methods:
  * Condoms (male or female) with or without a spermicide,
  * Diaphragm or cervical cap with spermicide,
  * Intrauterine device (IUD),
  * Hormonal contraception, or
  * Any other contraceptive method approved by the HVTN 124 Protocol Safety Review Team (PSRT)
  * Successful vasectomy in the male partner (considered successful if a volunteer reports that a male partner has [1] documentation of azoospermia by microscopy, or [2] a vasectomy more than 2 years ago with no resultant pregnancy despite sexual activity postvasectomy);
  * Or not be of reproductive potential, such as having reached menopause (no menses for 1 year) or having undergone hysterectomy, bilateral oophorectomy, or tubal ligation;
  * Or be sexually abstinent.
* Volunteers who were born female must also agree not to seek pregnancy through alternative methods, such as artificial insemination or in vitro fertilization until after the last required protocol clinic visit

Exclusion Criteria:

General

* Blood products received within 120 days before first vaccination
* Investigational research agents received within 30 days before first vaccination
* Body mass index (BMI) greater than or equal to 40; or BMI greater than or equal to 35 with 2 or more of the following: age greater than 45, systolic blood pressure greater than 140 mm Hg, diastolic blood pressure greater than 90 mm Hg, current smoker, known hyperlipidemia
* Intent to participate in another study of an investigational research agent or any other study that requires non-HVTN HIV antibody testing during the planned duration of the HVTN 124 study
* Pregnant or breastfeeding
* Active duty and reserve US military personnel

Vaccines and other Injections

* HIV vaccine(s) received in a prior HIV vaccine trial. For volunteers who have received control/placebo in an HIV vaccine trial, the HVTN 124 PSRT will determine eligibility on a case-by-case basis.
* Non-HIV experimental vaccine(s) received within the last 5 years in a prior vaccine trial. Exceptions may be made by the HVTN 124 PSRT for vaccines that have subsequently undergone licensure by the FDA. For volunteers who have received control/placebo in an experimental vaccine trial, the HVTN 124 PSRT will determine eligibility on a case-by-case basis. For volunteers who have received an experimental vaccine(s) greater than 5 years ago, eligibility for enrollment will be determined by the HVTN 124 PSRT on a case-by-case basis.
* Live attenuated vaccines received within 30 days before first vaccination or scheduled within 14 days after injection (eg, measles, mumps, and rubella [MMR]; oral polio vaccine [OPV]; varicella; yellow fever)
* Any vaccines that are not live attenuated vaccines and were received within 14 days prior to first vaccination (eg, tetanus, pneumococcal, Hepatitis A or B)
* Allergy treatment with antigen injections within 30 days before first vaccination or that are scheduled within 14 days after first vaccination

Immune System

* Immunosuppressive medications received within 168 days before first vaccination (Not exclusionary: [1] corticosteroid nasal spray; [2] inhaled corticosteroids; [3] topical corticosteroids for mild, uncomplicated dermatitis; or [4] a single course of oral/parenteral prednisone or equivalent at doses less than 60 mg/day and length of therapy less than 11 days with completion at least 30 days prior to enrollment.)
* Serious adverse reactions to vaccines or to vaccine components including history of anaphylaxis and related symptoms such as hives, respiratory difficulty, angioedema, and/or abdominal pain. (Not excluded from participation: a volunteer who had a nonanaphylactic adverse reaction to pertussis vaccine as a child.)
* Immunoglobulin received within 60 days before first vaccination
* Autoimmune disease, connective tissue disease, or history of vasculitis, e.g., leukocytoclastic vasculitis, Henoch-Schonlein purpura
* Immunodeficiency

Clinically significant medical conditions

* Untreated or incompletely treated syphilis infection
* Clinically significant medical condition, physical examination findings, clinically significant abnormal laboratory results, or past medical history with clinically significant implications for current health. A clinically significant condition or process includes but is not limited to:

  * A process that would affect the immune response,
  * A process that would require medication that affects the immune response,
  * Any contraindication to repeated injections or blood draws,
  * A condition that requires active medical intervention or monitoring to avert grave danger to the volunteer's health or well-being during the study period,
  * A condition or process for which signs or symptoms could be confused with reactions to vaccine, or
  * Any condition specifically listed among the exclusion criteria below.
* Any medical, psychiatric, occupational, or other condition that, in the judgment of the investigator, would interfere with, or serve as a contraindication to, protocol adherence, assessment of safety or reactogenicity, or a volunteer's ability to give informed consent
* Psychiatric condition that precludes compliance with the protocol. Specifically excluded are persons with psychoses within the past 3 years, ongoing risk for suicide, or history of suicide attempt or gesture within the past 3 years.
* Current anti-tuberculosis (TB) prophylaxis or therapy
* Asthma exclusion criteria: Asthma other than mild, well-controlled asthma. (Symptoms of asthma severity as defined in the most recent National Asthma Education and Prevention Program (NAEPP) Expert Panel report). Exclude a volunteer who:

  * Uses a short-acting rescue inhaler (typically a beta 2 agonist) daily, or
  * Uses moderate/high dose inhaled corticosteroids, or
  * In the past year has either of the following:
  * Greater than 1 exacerbation of symptoms treated with oral/parenteral corticosteroids;
  * Needed emergency care, urgent care, hospitalization, or intubation for asthma.
* Diabetes mellitus type 1 or type 2, including cases controlled with diet alone. (Not excluded: history of isolated gestational diabetes.)
* Thyroidectomy, or thyroid disease requiring medication during the last 12 months
* Hypertension:

  * If a person has been found to have elevated blood pressure or hypertension during screening or previously, exclude for blood pressure that is not well controlled. Well-controlled blood pressure is defined as consistently less than or equal to 140 mm Hg systolic and less than or equal to 90 mm Hg diastolic, with or without medication, with only isolated, brief instances of higher readings, which must be less than or equal to 150 mm Hg systolic and less than or equal to 100 mm Hg diastolic. For these volunteers, blood pressure must be less than or equal to 140 mm Hg systolic and less than or equal to 90 mm Hg diastolic at enrollment.
  * If a person has NOT been found to have elevated blood pressure or hypertension during screening or previously, exclude for systolic blood pressure greater than or equal to 150 mm Hg at enrollment or diastolic blood pressure greater than or equal to 100 mm Hg at enrollment.
* Bleeding disorder diagnosed by a doctor (eg, factor deficiency, coagulopathy, or platelet disorder requiring special precautions)
* Malignancy (Not excluded from participation: Volunteer who has had malignancy excised surgically and who, in the investigator's estimation, has a reasonable assurance of sustained cure, or who is unlikely to experience recurrence of malignancy during the period of the study)
* Seizure disorder: History of seizure(s) within past three years. Also exclude if volunteer has used medications in order to prevent or treat seizure(s) at any time within the past 3 years.
* Asplenia: any condition resulting in the absence of a functional spleen
* History of hereditary angioedema, acquired angioedema, or idiopathic angioedema.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2018-03-16 (Actual); Primary Completion 2020-05-11 (Actual); Study Completion 2020-10-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ian Frank, Study Chair — University of Pennsylvania; Turner Overton, Study Chair — University of Alabama at Birmingham
Locations (6):
- United States (6):
  - Alabama CRS, Birmingham, Alabama
  - The Hope Clinic of the Emory Vaccine Center CRS, Decatur, Georgia
  - Fenway Health (FH) CRS, Boston, Massachusetts
  - University of Rochester Vaccines to Prevent HIV Infection CRS, Rochester, New York
  - Case Clinical Research Site, Cleveland, Ohio
  - Penn Prevention CRS, Philadelphia, Pennsylvania

REFERENCES:
- [Derived] Jamieson PJ, Shen X, Abu-Shmais AA, Wasdin PT, Janowska K, Edwards RJ, Scapellato G, Bukenya M, Bass LE, Richardson SI, Manamela NP, Liu S, Barr M, Adams L, Paola Velez-Castro C, McCarthy C, Alexander CA, Gillespie RA, Mimms J, Suryadevara N, Sornberger TA, Zost SJ, Parks R, Flaherty S, Janke AK, Howard BN, Suresh YP, Ruprecht RM, Crowe JE Jr, Carnahan RH, Bailey JR, Kanekiyo M, Lingwood D, Haynes BF, Moore PL, Bonami RH, Tomaras GD, Archarya P, Montefiori DC, Kalams SA, Lu S, Georgiev IS. Glycan-reactive antibodies isolated from human HIV-1 vaccine trial participants show broad pathogen cross-reactivity. J Virol. 2025 Dec 23;99(12):e0125625. doi: 10.1128/jvi.01256-25. Epub 2025 Nov 10. PMID 41212034
- [Derived] Moodie Z, Li SS, Giorgi EE, Williams LD, Dintwe O, Carpp LN, Chen S, Seaton KE, Sawant SS, Zhang L, Heptinstall J, Liu S, Grunenberg N, Tomaka F, Rerks-Ngarm S, Pitisuttithum P, Nitayaphan S, Ake JA, Vasan S, Pantaleo G, Frank I, Baden LR, Goepfert PA, Keefer M, Chirenje M, Hosseinipour MC, Mngadi K, Laher F, Garrett N, Bekker LG, De Rosa S, Andersen-Nissen E, Kublin JG, Lu S, Gilbert PB, Gray GE, Corey L, McElrath MJ, Tomaras GD. A polyvalent DNA prime with matched polyvalent protein/GLA-SE boost regimen elicited the most robust and broad IgG and IgG3 V1V2 binding antibody and CD4+ T cell responses among 13 HIV vaccine trials. Emerg Microbes Infect. 2025 Dec;14(1):2485317. doi: 10.1080/22221751.2025.2485317. Epub 2025 Apr 7. PMID 40190112
- [Derived] Frank I, Li SS, Grunenberg N, Overton ET, Robinson ST, Zheng H, Seaton KE, Heptinstall JR, Allen MA, Mayer KH, Culver DA, Keefer MC, Edupuganti S, Pensiero MN, Mehra VL, De Rosa SC, Morris DE, Wang S, Seaman MS, Montefiori DC, Ferrari G, Tomaras GD, Kublin JG, Corey L, Lu S; HVTN 124 Study Team. Safety and immunogenicity of a polyvalent DNA-protein HIV vaccine with matched Env immunogens delivered as a prime-boost regimen or coadministered in HIV-uninfected adults in the USA (HVTN 124): a phase 1, placebo-controlled, double-blind randomised controlled trial. Lancet HIV. 2024 May;11(5):e285-e299. doi: 10.1016/S2352-3018(24)00036-5. PMID 38692824

RESULTS

PARTICIPANT FLOW:
Groups:
- Part A: Placebo: Placebo: Sodium Chloride USP 0.9% at Month (0, 2)
- Part A: Vaccine: Protein/ GLA-SE at Month (0, 2)
- Part B: Placebo: Placebo: Sodium Chloride USP 0.9% at Month (0, 1, 3, 6, 8)
- Part B: Vaccine 1: DNA+Placebo for protein at Month(0, 1, 3), Protein/GLA-SE+Placebo for DNA at Month (6, 8)
- Part B: Vaccine 2: DNA+Protein/GLA-SE at Month (0, 1, 3, 6, 8)
Period: Overall Study
Arm/Group | Part A: Placebo | Part A: Vaccine | Part B: Placebo | Part B: Vaccine 1 | Part B: Vaccine 2
Started | 2 | 10 | 6 | 21 | 21
Month 2.5 Immunogenicity Cohort | 2 | 10 | 0 | 0 | 0
Month 8.5 Immunogenicity Cohort | 0 | 0 | 6 | 19 | 16
Completed | 2 | 10 | 6 | 19 | 18
Not Completed | 0 | 0 | 0 | 2 | 3
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A: Placebo | Part A: Vaccine | Part B: Placebo | Part B: Vaccine 1 | Part B: Vaccine 2 | Total
Number analyzed (Participants) | 2 | 10 | 6 | 21 | 21 | 60
Age, Continuous [Median (Full Range); unit: years] | 36.5 [26 to 47] | 22.5 [18 to 47] | 29 [27 to 36] | 25 [19 to 40] | 31 [21 to 48] | 26.5 [18 to 48]
Age, Customized [Count of Participants; unit: Participants]
  Less than 18 years | 0 | 0 | 0 | 0 | 0 | 0
  18 - 20 years | 0 | 4 | 0 | 3 | 0 | 7
  21 - 30 years | 1 | 3 | 4 | 12 | 10 | 30
  31 - 40 years | 0 | 1 | 2 | 6 | 9 | 18
  41 - 50 years | 1 | 2 | 0 | 0 | 2 | 5
  Above 50 years | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 6 | 3 | 13 | 11 | 34
  Male | 1 | 4 | 3 | 8 | 10 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 1 | 1 | 2
  Not Hispanic or Latino | 2 | 10 | 6 | 20 | 20 | 58
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 2 | 0 | 2 | 2 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 1 | 3 | 0 | 5
  White | 1 | 7 | 4 | 14 | 17 | 43
  More than one race | 0 | 1 | 1 | 2 | 1 | 5
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  USA | 2 | 10 | 6 | 21 | 21 | 60

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting Local Reactogenicity Signs and Symptoms
Description: Graded according to the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events, Corrected Version 2.1, July 2017. The maximum grade observed for each symptom over the time frame is presented.
Time Frame: Measured through 3 days after participants' each vaccination at Months 0, 2 for part A and Months 0, 1, 3, 6, 8 for part B
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Placebo | Part A: Vaccine | Part B: Placebo | Part B: Vaccine 1 | Part B: Vaccine 2
Number analyzed (Participants) | 2 | 10 | 6 | 21 | 21
Participants
  Pain: None | 2 | 5 | 5 | 3 | 1
  Pain: Mild | 0 | 4 | 1 | 12 | 15
  Pain: Moderate | 0 | 1 | 0 | 5 | 4
  Pain: Severe | 0 | 0 | 0 | 1 | 1
  Pain: Potentially Life-threatening | 0 | 0 | 0 | 0 | 0
  Tenderness: None | 2 | 3 | 4 | 1 | 0
  Tenderness: Mild | 0 | 6 | 2 | 15 | 17
  Tenderness: Moderate | 0 | 1 | 0 | 4 | 3
  Tenderness: Severe | 0 | 0 | 0 | 1 | 1
  Tenderness: Potentially Life-threatening | 0 | 0 | 0 | 0 | 0
  Pain and/or Tenderness: None | 2 | 3 | 4 | 1 | 0
  Pain and/or Tenderness: Mild | 0 | 6 | 2 | 13 | 15
  Pain and/or Tenderness: Moderate | 0 | 1 | 0 | 6 | 5
  Pain and/or Tenderness: Severe | 0 | 0 | 0 | 1 | 1
  Pain and/or Tenderness: Potentially Life-threatening | 0 | 0 | 0 | 0 | 0
  Erythema: None | 2 | 10 | 6 | 14 | 13
  Erythema: Mild | 0 | 0 | 0 | 0 | 2
  Erythema: Moderate | 0 | 0 | 0 | 2 | 4
  Erythema: Severe | 0 | 0 | 0 | 5 | 2
  Erythema: Potentially Life-threatening | 0 | 0 | 0 | 0 | 0
  Induration: None | 2 | 10 | 6 | 16 | 14
  Induration: Mild | 0 | 0 | 0 | 1 | 3
  Induration: Moderate | 0 | 0 | 0 | 0 | 2
  Induration: Severe | 0 | 0 | 0 | 4 | 2
  Induration: Potentially Life-threatening | 0 | 0 | 0 | 0 | 0
  Erythema and/or Induration: None | 2 | 10 | 6 | 14 | 12
  Erythema and/or Induration: Mild | 0 | 0 | 0 | 0 | 3
  Erythema and/or Induration: Moderate | 0 | 0 | 0 | 2 | 4
  Erythema and/or Induration: Severe | 0 | 0 | 0 | 5 | 2
  Erythema and/or Induration: Potentially Life-threatening | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants Reporting Systemic Reactogenicity Signs and Symptoms
Description: as for outcome 1
Time Frame: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Placebo | Part A: Vaccine | Part B: Placebo | Part B: Vaccine 1 | Part B: Vaccine 2
Number analyzed (Participants) | 2 | 10 | 6 | 21 | 21
Participants
  Malaise and/or fatigue: None | 1 | 5 | 2 | 4 | 6
  Malaise and/or fatigue: Mild | 1 | 5 | 1 | 8 | 8
  Malaise and/or fatigue: Moderate | 0 | 0 | 2 | 7 | 6
  Malaise and/or fatigue: Severe | 0 | 0 | 1 | 2 | 1
  Malaise and/or fatigue: Potentially Life-threatening | 0 | 0 | 0 | 0 | 0
  Myalgia: None | 1 | 6 | 4 | 8 | 11
  Myalgia: Mild | 1 | 4 | 2 | 9 | 7
  Myalgia: Moderate | 0 | 0 | 0 | 2 | 1
  Myalgia: Severe | 0 | 0 | 0 | 2 | 2
  Myalgia: Potentially Life-threatening | 0 | 0 | 0 | 0 | 0
  Headache: None | 1 | 5 | 2 | 3 | 9
  Headache: Mild | 1 | 5 | 3 | 10 | 8
  Headache: Moderate | 0 | 0 | 1 | 8 | 2
  Headache: Severe | 0 | 0 | 0 | 0 | 2
  Headache: Potentially Life-threatening | 0 | 0 | 0 | 0 | 0
  Nausea: None | 1 | 8 | 4 | 12 | 15
  Nausea: Mild | 1 | 2 | 1 | 6 | 4
  Nausea: Moderate | 0 | 0 | 1 | 3 | 2
  Nausea: Severe | 0 | 0 | 0 | 0 | 0
  Nausea: Potentially Life-threatening | 0 | 0 | 0 | 0 | 0
  Vomiting: None | 2 | 10 | 6 | 17 | 18
  Vomiting: Mild | 0 | 0 | 0 | 3 | 1
  Vomiting: Moderate | 0 | 0 | 0 | 1 | 2
  Vomiting: Severe | 0 | 0 | 0 | 0 | 0
  Vomiting: Potentially Life-threatening | 0 | 0 | 0 | 0 | 0
  Chills: None | 2 | 10 | 6 | 11 | 15
  Chills: Mild | 0 | 0 | 0 | 4 | 4
  Chills: Moderate | 0 | 0 | 0 | 4 | 0
  Chills: Severe | 0 | 0 | 0 | 2 | 2
  Chills: Potentially Life-threatening | 0 | 0 | 0 | 0 | 0
  Arthralgia: None | 2 | 8 | 6 | 10 | 17
  Arthralgia: Mild | 0 | 1 | 0 | 8 | 2
  Arthralgia: Moderate | 0 | 1 | 0 | 1 | 1
  Arthralgia: Severe | 0 | 0 | 0 | 2 | 1
  Arthralgia: Potentially Life-threatening | 0 | 0 | 0 | 0 | 0
  Max. Systemic Symptoms: None | 1 | 3 | 2 | 3 | 5
  Max. Systemic Symptoms: Mild | 1 | 6 | 0 | 8 | 8
  Max. Systemic Symptoms: Moderate | 0 | 1 | 3 | 8 | 6
  Max. Systemic Symptoms: Severe | 0 | 0 | 1 | 2 | 2
  Max. Systemic Symptoms: Potentially Life-threatening | 0 | 0 | 0 | 0 | 0
  Temperature: None | 2 | 10 | 6 | 15 | 16
  Temperature: Mild | 0 | 0 | 0 | 2 | 3
  Temperature: Moderate | 0 | 0 | 0 | 3 | 2
  Temperature: Severe | 0 | 0 | 0 | 0 | 0
  Temperature: Potentially Life-threatening | 0 | 0 | 0 | 1 | 0

3. Primary Outcome: Number of Participants Reporting Adverse Events (AEs), by Relationship to Study Product
Description: For participants reporting multiple AEs over the time frame, the maximum relationship is counted.
Time Frame: Measured through 30 days after each vaccine dose at Months 0, 2 for part A and Months 0, 1, 3, 6, 8 for part B
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Placebo | Part A: Vaccine | Part B: Placebo | Part B: Vaccine 1 | Part B: Vaccine 2
Number analyzed (Participants) | 2 | 10 | 6 | 21 | 21
Participants
  Related | 0 | 0 | 0 | 5 | 2
  Not Related | 2 | 6 | 5 | 14 | 16
  No AE reported | 0 | 4 | 1 | 2 | 3

4. Primary Outcome: Number of Participants Reporting Adverse Events (AEs), by Severity Grade
Description: For participants reporting multiple AEs over the time frame, the maximum severity grade is counted.
Time Frame: Measured through 30 days after each vaccine dose at Months 0, 2 for part A and Months 0, 1, 3, 6, 8 for part B
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Placebo | Part A: Vaccine | Part B: Placebo | Part B: Vaccine 1 | Part B: Vaccine 2
Number analyzed (Participants) | 2 | 10 | 6 | 21 | 21
Participants
  Mild | 0 | 2 | 1 | 0 | 2
  Moderate | 2 | 4 | 4 | 18 | 14
  Severe | 0 | 0 | 0 | 1 | 2
  No AE reported | 0 | 4 | 1 | 2 | 3

5. Primary Outcome: Number of Participants Reporting Serious Adverse Events (SAEs)
Description: Measured as outlined in Version 2.0 (January 2010) of the Manual for Expedited Reporting of Adverse Events to DAIDS (DAIDS EAE Manual).
Time Frame: Measured through Month 8 for part A and Month 14 for part B
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Placebo | Part A: Vaccine | Part B: Placebo | Part B: Vaccine 1 | Part B: Vaccine 2
Number analyzed (Participants) | 2 | 10 | 6 | 21 | 21
Participants | 0 | 0 | 0 | 0 | 0

6. Primary Outcome: Number of Participants Reporting Adverse Events of Special Interest (AESIs)
Description: Adverse events of special interest were described in Appendix N of the protocol. AESI for this protocol include but are not limited to potential immune-mediated diseases. There were no adverse events of special interest reported by any participant.
Time Frame: Measured through Month 8 for part A and Month 14 for part B
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Placebo | Part A: Vaccine | Part B: Placebo | Part B: Vaccine 1 | Part B: Vaccine 2
Number analyzed (Participants) | 2 | 10 | 6 | 21 | 21
Participants | 0 | 0 | 0 | 0 | 0

7. Primary Outcome: Numbers of Participants With Grade 1 or Higher Local Laboratory Results
Description: The number (percentage) of participants with local laboratory values recorded as meeting Grade 1 AE criteria or above as specified in the DAIDS AE Grading Table were tabulated by treatment arm for each post-vaccination time point. Laboratory results are summarized by analyte and timepoint. Analytes and timepoint combinations with no grade 1 or higher results are not shown.
Time Frame: Measured during Screening, Day 14, Day 70, Day140 for part A and visits Screening, Day 14, Day 42, Day 98, Day 182, Day 238 and Day 334 for part B
Population: The "overall number of participants analyzed" represents participants enrolled and eligible for laboratory assessment. Participants do not have laboratory assessments if they attended the visit but laboratory specimens were not collected, or they missed the scheduled visit, or they terminated participation in the study prior to the scheduled visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Placebo | Part A: Vaccine | Part B: Placebo | Part B: Vaccine 1 | Part B: Vaccine 2
Number analyzed (Participants) | 2 | 10 | 6 | 21 | 21
Participants
  AST (U/L)- Day42: number analyzed (Participants) | 0 | 0 | 6 | 21 | 21
  AST (U/L)- Day42 |  |  | 0 | 1 | 0
  AST (U/L)- Day98: number analyzed (Participants) | 0 | 0 | 6 | 21 | 19
  AST (U/L)- Day98 |  |  | 0 | 0 | 1
  AST (U/L)- Day140: number analyzed (Participants) | 2 | 10 | 0 | 0 | 0
  AST (U/L)- Day140 | 0 | 1 |  |  |
  ALT (SGPT) (U/L)- Day42: number analyzed (Participants) | 0 | 0 | 6 | 21 | 21
  ALT (SGPT) (U/L)- Day42 |  |  | 0 | 1 | 0
  Hemoglobin (g/dL)- Day182: number analyzed (Participants) | 0 | 0 | 6 | 17 | 21
  Hemoglobin (g/dL)- Day182 |  |  | 0 | 2 | 0
  Hemoglobin (g/dL)- Day238: number analyzed (Participants) | 0 | 0 | 6 | 18 | 21
  Hemoglobin (g/dL)- Day238 |  |  | 0 | 1 | 0
  Hemoglobin (g/dL)- Day334: number analyzed (Participants) | 0 | 0 | 6 | 18 | 21
  Hemoglobin (g/dL)- Day334 |  |  | 0 | 1 | 0
  Creatinine (g/dL)- Day14 | 0 | 2 | 0 | 0 | 0
  Creatinine (g/dL)- Day42: number analyzed (Participants) | 0 | 0 | 6 | 21 | 19
  Creatinine (g/dL)- Day42 |  |  | 0 | 0 | 1
  Creatinine (g/dL)- Day98: number analyzed (Participants) | 0 | 0 | 6 | 19 | 21
  Creatinine (g/dL)- Day98 |  |  | 0 | 2 | 0
  Creatinine (g/dL)- Day182: number analyzed (Participants) | 0 | 0 | 6 | 17 | 18
  Creatinine (g/dL)- Day182 |  |  | 0 | 2 | 2
  Creatinine (g/dL)- Day334: number analyzed (Participants) | 0 | 0 | 6 | 21 | 16
  Creatinine (g/dL)- Day334 |  |  | 1 | 0 | 1

8. Primary Outcome: Alk Phos, AST, ALT in UL
Description: Laboratory results are summarized by analyte and timepoint.
Time Frame: Measured through Screening, Day 14, Day 70, Day140 for part A and visits Screening, Day 14, Day 42, Day 98, Day 182, Day 238 and Day 334 for part B
Population: as for outcome 7
Measure: Median (Inter-Quartile Range); unit: U/L
Arm/Group | Part A: Placebo | Part A: Vaccine | Part B: Placebo | Part B: Vaccine 1 | Part B: Vaccine 2
Number analyzed (Participants) | 2 | 10 | 6 | 21 | 21
U/L
  Alkaline Phosphatase (U/L)- Screening | 61 [58 to 64] | 59.5 [46 to 69] | 54.5 [51 to 60] | 61 [56 to 74] | 59 [52 to 78]
  Alkaline Phosphatase (U/L)- Day14: number analyzed (Participants) | 2 | 10 | 6 | 21 | 20
  Alkaline Phosphatase (U/L)- Day14 | 57.5 [46 to 69] | 56 [43 to 81] | 53 [49 to 56] | 62 [56 to 71] | 60 [51 to 65.5]
  Alkaline Phosphatase (U/L)- Day42: number analyzed (Participants) | 0 | 0 | 6 | 21 | 19
  Alkaline Phosphatase (U/L)- Day42 |  |  | 56 [53 to 59] | 69 [58 to 73] | 57 [51 to 68]
  Alkaline Phosphatase (U/L)- Day70: number analyzed (Participants) | 2 | 10 | 0 | 0 | 0
  Alkaline Phosphatase (U/L)- Day70 | 54 [51 to 57] | 55 [50 to 76] |  |  |
  Alkaline Phosphatase (U/L)- Day98: number analyzed (Participants) | 0 | 0 | 5 | 19 | 19
  Alkaline Phosphatase (U/L)- Day98 |  |  | 54 [51 to 57] | 64 [54 to 77] | 61 [50 to 72]
  Alkaline Phosphatase (U/L)- Day140: number analyzed (Participants) | 2 | 10 | 0 | 0 | 0
  Alkaline Phosphatase (U/L)- Day140 | 57.5 [50 to 65] | 59 [50 to 68] |  |  |
  Alkaline Phosphatase (U/L)- Day182: number analyzed (Participants) | 0 | 0 | 6 | 17 | 18
  Alkaline Phosphatase (U/L)- Day182 |  |  | 59.5 [52 to 61] | 63 [56 to 72] | 60.5 [44 to 68]
  Alkaline Phosphatase (U/L)- Day238: number analyzed (Participants) | 0 | 0 | 6 | 18 | 16
  Alkaline Phosphatase (U/L)- Day238 |  |  | 52 [50 to 73] | 61.5 [52 to 72] | 58.5 [49 to 69]
  Alkaline Phosphatase (U/L)- Day334: number analyzed (Participants) | 0 | 0 | 6 | 18 | 16
  Alkaline Phosphatase (U/L)- Day334 |  |  | 52.5 [50 to 67] | 62.5 [52 to 66] | 62 [50 to 67.5]
  AST (U/L)- Screening | 18 [16 to 20] | 19 [16 to 19] | 16.5 [15 to 27] | 16 [14 to 19] | 19 [18 to 23]
  AST (U/L)- Day14: number analyzed (Participants) | 2 | 10 | 6 | 21 | 20
  AST (U/L)- Day14 | 19 [16 to 22] | 15 [14 to 19] | 19.5 [18 to 25] | 17 [14 to 20] | 19 [16 to 20]
  AST (U/L)- Day42: number analyzed (Participants) | 0 | 0 | 6 | 21 | 19
  AST (U/L)- Day42 |  |  | 17 [13 to 20] | 15 [15 to 21] | 17 [16 to 20]
  AST (U/L)- Day70: number analyzed (Participants) | 2 | 10 | 0 | 0 | 0
  AST (U/L)- Day70 | 13 [12 to 14] | 17 [15 to 19] |  |  |
  AST (U/L)- Day98: number analyzed (Participants) | 0 | 0 | 5 | 19 | 19
  AST (U/L)- Day98 |  |  | 16 [16 to 20] | 17 [14 to 20] | 18 [16 to 21]
  AST (U/L)- Day140: number analyzed (Participants) | 2 | 10 | 0 | 0 | 0
  AST (U/L)- Day140 | 13.5 [12 to 15] | 17 [15 to 26] |  |  |
  AST (U/L)- Day182: number analyzed (Participants) | 0 | 0 | 6 | 17 | 18
  AST (U/L)- Day182 |  |  | 14.5 [12 to 16] | 16 [15 to 18] | 17.5 [16 to 18]
  AST (U/L)- Day238: number analyzed (Participants) | 0 | 0 | 6 | 18 | 16
  AST (U/L)- Day238 |  |  | 15.5 [13 to 18] | 16 [14 to 18] | 16 [15.5 to 22]
  AST (U/L)- Day334: number analyzed (Participants) | 0 | 0 | 6 | 18 | 16
  AST (U/L)- Day334 |  |  | 15.5 [14 to 24] | 16 [14 to 18] | 19 [15.5 to 21]
  ALT (SGPT) (U/L)- Screening | 22 [21 to 23] | 14.5 [11 to 21] | 22.5 [16 to 25] | 13 [10 to 18] | 16 [13 to 24]
  ALT (SGPT) (U/L)- Day14: number analyzed (Participants) | 2 | 10 | 6 | 21 | 20
  ALT (SGPT) (U/L)- Day14 | 21.5 [19 to 24] | 10 [8 to 19] | 19.5 [16 to 30] | 14 [12 to 18] | 15 [12.5 to 20.5]
  ALT (SGPT) (U/L)- Day42: number analyzed (Participants) | 0 | 0 | 6 | 21 | 19
  ALT (SGPT) (U/L)- Day42 |  |  | 17 [12 to 20] | 14 [11 to 16] | 15 [11 to 22]
  ALT (SGPT) (U/L)- Day70: number analyzed (Participants) | 2 | 10 | 0 | 0 | 0
  ALT (SGPT) (U/L)- Day70 | 18 [11 to 25] | 14.5 [10 to 19] |  |  |
  ALT (SGPT) (U/L)- Day98: number analyzed (Participants) | 0 | 0 | 5 | 19 | 19
  ALT (SGPT) (U/L)- Day98 |  |  | 15 [15 to 16] | 14 [11 to 17] | 15 [10 to 19]
  ALT (SGPT) (U/L)- Day140: number analyzed (Participants) | 2 | 10 | 0 | 0 | 0
  ALT (SGPT) (U/L)- Day140 | 21 [11 to 31] | 14.5 [12 to 20] |  |  |
  ALT (SGPT) (U/L)- Day182: number analyzed (Participants) | 0 | 0 | 6 | 17 | 18
  ALT (SGPT) (U/L)- Day182 |  |  | 12.5 [10 to 19] | 12 [10 to 15] | 15.5 [14 to 19]
  ALT (SGPT) (U/L)- Day238: number analyzed (Participants) | 0 | 0 | 6 | 18 | 16
  ALT (SGPT) (U/L)- Day238 |  |  | 15.5 [11 to 19] | 11.5 [11 to 15] | 12.5 [9 to 22]
  ALT (SGPT) (U/L)- Day334: number analyzed (Participants) | 0 | 0 | 6 | 18 | 16
  ALT (SGPT) (U/L)- Day334 |  |  | 17 [12 to 20] | 13 [10 to 15] | 15.5 [12 to 26.5]

9. Primary Outcome: Hemoglobin, Creatinine in g/dL
Description: Laboratory results are summarized by analyte and timepoint.
Time Frame: as for outcome 8
Population: as for outcome 7
Measure: Median (Inter-Quartile Range); unit: g/dL
Arm/Group | Part A: Placebo | Part A: Vaccine | Part B: Placebo | Part B: Vaccine 1 | Part B: Vaccine 2
Number analyzed (Participants) | 2 | 10 | 6 | 21 | 21
g/dL
  Hemoglobin (g/dL)- Screening | 14.7 [13.7 to 15.7] | 13.75 [12.7 to 15.2] | 13.85 [13.2 to 14.6] | 14.7 [13.2 to 15] | 14.8 [13.4 to 15.4]
  Hemoglobin (g/dL)- Day14: number analyzed (Participants) | 2 | 10 | 6 | 21 | 20
  Hemoglobin (g/dL)- Day14 | 14.65 [14.4 to 14.9] | 13.45 [12.8 to 14.3] | 13.5 [12.3 to 14.4] | 13.5 [12.5 to 14.8] | 13.95 [12.75 to 14.7]
  Hemoglobin (g/dL)- Day42: number analyzed (Participants) | 0 | 0 | 6 | 21 | 19
  Hemoglobin (g/dL)- Day42 |  |  | 13.9 [12.5 to 14.4] | 13.8 [13.1 to 14.5] | 13.8 [13.3 to 15.1]
  Hemoglobin (g/dL)- Day70: number analyzed (Participants) | 2 | 10 | 0 | 0 | 0
  Hemoglobin (g/dL)- Day70 | 13.25 [12.5 to 14] | 14.1 [13 to 14.5] |  |  |
  Hemoglobin (g/dL)- Day98: number analyzed (Participants) | 0 | 0 | 5 | 19 | 19
  Hemoglobin (g/dL)- Day98 |  |  | 13.2 [12.7 to 14.6] | 14 [12.9 to 14.7] | 14.8 [13.4 to 15.3]
  Hemoglobin (g/dL)- Day140: number analyzed (Participants) | 2 | 10 | 0 | 0 | 0
  Hemoglobin (g/dL)- Day140 | 14.35 [13 to 15.7] | 13.65 [12.3 to 14.6] |  |  |
  Hemoglobin (g/dL)- Day182: number analyzed (Participants) | 0 | 0 | 6 | 17 | 18
  Hemoglobin (g/dL)- Day182 |  |  | 13.6 [12.2 to 14] | 13.4 [11.6 to 14.2] | 14 [13.2 to 14.8]
  Hemoglobin (g/dL)- Day238: number analyzed (Participants) | 0 | 0 | 6 | 18 | 16
  Hemoglobin (g/dL)- Day238 |  |  | 13.5 [11.2 to 14.4] | 13.2 [12.2 to 14] | 14 [12.8 to 15.1]
  Hemoglobin (g/dL)- Day334: number analyzed (Participants) | 0 | 0 | 6 | 18 | 16
  Hemoglobin (g/dL)- Day334 |  |  | 14.25 [11.4 to 14.6] | 12.75 [12.1 to 14.3] | 14.15 [13.25 to 14.85]
  Creatinine (g/dL)- Screening | 0.00094 [0.00079 to 0.00109] | 0.00077 [0.00068 to 0.00093] | 0.000795 [0.00074 to 0.00091] | 0.00078 [0.00068 to 0.00083] | 0.0008 [0.00075 to 0.0009]
  Creatinine (g/dL)- Day14: number analyzed (Participants) | 2 | 10 | 6 | 21 | 20
  Creatinine (g/dL)- Day14 | 0.00102 [0.0008 to 0.00124] | 0.000815 [0.00079 to 0.00092] | 0.000835 [0.00077 to 0.00093] | 0.00075 [0.00071 to 0.00085] | 0.000835 [0.00075 to 0.00091]
  Creatinine (g/dL)- Day42: number analyzed (Participants) | 0 | 0 | 6 | 21 | 19
  Creatinine (g/dL)- Day42 |  |  | 0.00081 [0.00071 to 0.00099] | 0.00079 [0.00071 to 0.00083] | 0.00087 [0.00073 to 0.00094]
  Creatinine (g/dL)- Day70: number analyzed (Participants) | 2 | 10 | 0 | 0 | 0
  Creatinine (g/dL)- Day70 | 0.00088 [0.00072 to 0.00104] | 0.00075 [0.0007 to 0.00096] |  |  |
  Creatinine (g/dL)- Day98: number analyzed (Participants) | 0 | 0 | 5 | 19 | 19
  Creatinine (g/dL)- Day98 |  |  | 0.00083 [0.00075 to 0.0009] | 0.0008 [0.0007 to 0.00086] | 0.00084 [0.00075 to 0.001]
  Creatinine (g/dL)- Day140: number analyzed (Participants) | 2 | 10 | 0 | 0 | 0
  Creatinine (g/dL)- Day140 | 0.000935 [0.00086 to 0.00101] | 0.000765 [0.00069 to 0.00095] |  |  |
  Creatinine (g/dL)- Day182: number analyzed (Participants) | 0 | 0 | 6 | 17 | 18
  Creatinine (g/dL)- Day182 |  |  | 0.00085 [0.00072 to 0.00092] | 0.00088 [0.00078 to 0.00094] | 0.000855 [0.0008 to 0.00105]
  Creatinine (g/dL)- Day238: number analyzed (Participants) | 0 | 0 | 6 | 18 | 16
  Creatinine (g/dL)- Day238 |  |  | 0.000815 [0.00076 to 0.00087] | 0.00076 [0.0007 to 0.00082] | 0.000845 [0.00076 to 0.00092]
  Creatinine (g/dL)- Day334: number analyzed (Participants) | 0 | 0 | 6 | 18 | 16
  Creatinine (g/dL)- Day334 |  |  | 0.00082 [0.00076 to 0.00104] | 0.00081 [0.0007 to 0.00088] | 0.000895 [0.0008 to 0.00097]

10. Primary Outcome: WBC, Platelets, Lymphocytes, Neutrophils in Thousand Cells/Cubic mm
Description: Laboratory results are summarized by analyte and timepoint.
Time Frame: as for outcome 8
Population: as for outcome 7
Measure: Median (Inter-Quartile Range); unit: thousand cells/cubic mm
Arm/Group | Part A: Placebo | Part A: Vaccine | Part B: Placebo | Part B: Vaccine 1 | Part B: Vaccine 2
Number analyzed (Participants) | 2 | 10 | 6 | 21 | 21
thousand cells/cubic mm
  WBC (1000/cubic mm)- Screening | 5.1 [4.4 to 5.8] | 6.305 [4.8 to 7.3] | 5.9 [5.3 to 6.2] | 5.7 [5.2 to 7.1] | 6.4 [5.5 to 7.4]
  WBC (1000/cubic mm)- Day14: number analyzed (Participants) | 2 | 10 | 6 | 21 | 20
  WBC (1000/cubic mm)- Day14 | 4.35 [3.4 to 5.3] | 5.62 [4.4 to 7.5] | 5.65 [4.8 to 6.6] | 6 [5.6 to 6.8] | 6.4 [5.185 to 6.85]
  WBC (1000/cubic mm)- Day42: number analyzed (Participants) | 0 | 0 | 6 | 21 | 19
  WBC (1000/cubic mm)- Day42 |  |  | 6.45 [5.4 to 8.3] | 6.2 [5.1 to 7.1] | 6.3 [5.3 to 6.9]
  WBC (1000/cubic mm)- Day70: number analyzed (Participants) | 2 | 10 | 0 | 0 | 0
  WBC (1000/cubic mm)- Day70 | 5.8 [3.6 to 8] | 6.12 [5.6 to 7.3] |  |  |
  WBC (1000/cubic mm)- Day98: number analyzed (Participants) | 0 | 0 | 5 | 19 | 19
  WBC (1000/cubic mm)- Day98 |  |  | 5.8 [5.6 to 6] | 6.11 [5.3 to 7.1] | 5.7 [4.8 to 6.7]
  WBC (1000/cubic mm)- Day140: number analyzed (Participants) | 2 | 10 | 0 | 0 | 0
  WBC (1000/cubic mm)- Day140 | 4.15 [4.1 to 4.2] | 6.26 [4.9 to 9.1] |  |  |
  WBC (1000/cubic mm)- Day182: number analyzed (Participants) | 0 | 0 | 6 | 17 | 18
  WBC (1000/cubic mm)- Day182 |  |  | 6 [5.4 to 6.6] | 5.6 [5.1 to 7.1] | 6.25 [5 to 7]
  WBC (1000/cubic mm)- Day238: number analyzed (Participants) | 0 | 0 | 6 | 18 | 16
  WBC (1000/cubic mm)- Day238 |  |  | 6 [4.8 to 6.2] | 6 [5 to 7] | 6.15 [5.57 to 6.75]
  WBC (1000/cubic mm)- Day334: number analyzed (Participants) | 0 | 0 | 6 | 18 | 16
  WBC (1000/cubic mm)- Day334 |  |  | 5.4 [5 to 6.2] | 5.6 [5.01 to 6.7] | 5.88 [5.25 to 6.65]
  Platelets (1000/cubic mm)- Screening | 288 [236 to 340] | 296 [266.9 to 341] | 229 [217 to 387] | 250 [212 to 295] | 246 [210 to 273]
  Platelets (1000/cubic mm)- Day14: number analyzed (Participants) | 2 | 10 | 6 | 21 | 20
  Platelets (1000/cubic mm)- Day14 | 297 [205 to 389] | 297.5 [259 to 323] | 236 [210 to 328] | 244 [205 to 277] | 226.5 [201.55 to 278.5]
  Platelets (1000/cubic mm)- Day42: number analyzed (Participants) | 0 | 0 | 6 | 21 | 19
  Platelets (1000/cubic mm)- Day42 |  |  | 238 [207 to 334] | 243 [209 to 313] | 260.5 [193 to 291]
  Platelets (1000/cubic mm)- Day70: number analyzed (Participants) | 2 | 10 | 0 | 0 | 0
  Platelets (1000/cubic mm)- Day70 | 277.5 [243 to 312] | 286 [266 to 308] |  |  |
  Platelets (1000/cubic mm)- Day98: number analyzed (Participants) | 0 | 0 | 5 | 19 | 19
  Platelets (1000/cubic mm)- Day98 |  |  | 223 [203 to 256] | 244 [193 to 311] | 224 [191.1 to 268]
  Platelets (1000/cubic mm)- Day140: number analyzed (Participants) | 2 | 10 | 0 | 0 | 0
  Platelets (1000/cubic mm)- Day140 | 264.5 [243 to 286] | 287 [274 to 304] |  |  |
  Platelets (1000/cubic mm)- Day182: number analyzed (Participants) | 0 | 0 | 6 | 17 | 18
  Platelets (1000/cubic mm)- Day182 |  |  | 215.5 [205 to 328] | 278 [201 to 362.6] | 232 [190 to 287]
  Platelets (1000/cubic mm)- Day238: number analyzed (Participants) | 0 | 0 | 6 | 18 | 16
  Platelets (1000/cubic mm)- Day238 |  |  | 234.5 [210 to 315] | 266.1 [229 to 336] | 239.8 [188 to 287.9]
  Platelets (1000/cubic mm)- Day334: number analyzed (Participants) | 0 | 0 | 6 | 18 | 16
  Platelets (1000/cubic mm)- Day334 |  |  | 253.5 [197 to 339] | 280 [218 to 347] | 239.05 [192 to 273.5]
  Lymphocytes (1000/cubic mm)- Screening | 2.189 [1.148 to 3.23] | 1.942 [1.579 to 2.403] | 1.7635 [1.63 to 1.911] | 1.918 [1.664 to 2.213] | 2.134 [1.863 to 2.28]
  Lymphocytes (1000/cubic mm)- Day14: number analyzed (Participants) | 2 | 10 | 6 | 21 | 20
  Lymphocytes (1000/cubic mm)- Day14 | 2.037 [1.054 to 3.02] | 1.7895 [1.452 to 2.001] | 1.8115 [1.613 to 1.876] | 1.848 [1.56 to 2.237] | 1.935 [1.6725 to 2.1865]
  Lymphocytes (1000/cubic mm)- Day42: number analyzed (Participants) | 0 | 0 | 6 | 21 | 19
  Lymphocytes (1000/cubic mm)- Day42 |  |  | 1.583 [1.361 to 1.879] | 1.85 [1.415 to 2.313] | 1.93 [1.742 to 2.144]
  Lymphocytes (1000/cubic mm)- Day70: number analyzed (Participants) | 2 | 10 | 0 | 0 | 0
  Lymphocytes (1000/cubic mm)- Day70 | 2.0955 [1.051 to 3.14] | 2.1495 [1.712 to 2.467] |  |  |
  Lymphocytes (1000/cubic mm)- Day98: number analyzed (Participants) | 0 | 0 | 5 | 19 | 19
  Lymphocytes (1000/cubic mm)- Day98 |  |  | 1.589 [1.534 to 1.773] | 1.8 [1.461 to 2.081] | 1.98 [1.6 to 2.165]
  Lymphocytes (1000/cubic mm)- Day140: number analyzed (Participants) | 2 | 10 | 0 | 0 | 0
  Lymphocytes (1000/cubic mm)- Day140 | 1.574 [1.168 to 1.98] | 1.9625 [1.486 to 2.75] |  |  |
  Lymphocytes (1000/cubic mm)- Day182: number analyzed (Participants) | 0 | 0 | 6 | 17 | 18
  Lymphocytes (1000/cubic mm)- Day182 |  |  | 1.659 [1.507 to 1.822] | 2.076 [1.501 to 2.421] | 1.945 [1.591 to 2.19]
  Lymphocytes (1000/cubic mm)- Day238: number analyzed (Participants) | 0 | 0 | 6 | 18 | 16
  Lymphocytes (1000/cubic mm)- Day238 |  |  | 1.679 [1.535 to 1.959] | 1.928 [1.78 to 2.057] | 1.6865 [1.504 to 1.8315]
  Lymphocytes (1000/cubic mm)- Day334: number analyzed (Participants) | 0 | 0 | 6 | 18 | 16
  Lymphocytes (1000/cubic mm)- Day334 |  |  | 1.5425 [1.465 to 1.795] | 1.96 [1.48 to 2.25] | 1.745 [1.587 to 1.97]
  Neutrophils (1000/cubic mm)- Screening | 2.22 [1.862 to 2.578] | 3.848 [2.875 to 5.313] | 3.568 [3.403 to 3.837] | 3.648 [2.77 to 4.023] | 3.41 [2.965 to 4.788]
  Neutrophils (1000/cubic mm)- Day14: number analyzed (Participants) | 2 | 10 | 6 | 21 | 20
  Neutrophils (1000/cubic mm)- Day14 | 1.7345 [1.635 to 1.834] | 3.322 [2.411 to 5.1] | 3.2585 [2.41 to 4] | 3.397 [3.144 to 4.141] | 3.4945 [2.405 to 4.112]
  Neutrophils (1000/cubic mm)- Day42: number analyzed (Participants) | 0 | 0 | 6 | 21 | 19
  Neutrophils (1000/cubic mm)- Day42 |  |  | 3.7595 [3.375 to 6.01] | 3.66 [2.885 to 4.509] | 3.317 [2.945 to 3.95]
  Neutrophils (1000/cubic mm)- Day70: number analyzed (Participants) | 2 | 10 | 0 | 0 | 0
  Neutrophils (1000/cubic mm)- Day70 | 3.072 [1.904 to 4.24] | 3.9035 [3.161 to 4.417] |  |  |
  Neutrophils (1000/cubic mm)- Day98: number analyzed (Participants) | 0 | 0 | 5 | 19 | 19
  Neutrophils (1000/cubic mm)- Day98 |  |  | 3.492 [3.27 to 3.578] | 3.67 [2.749 to 4.303] | 3.101 [2.235 to 4.541]
  Neutrophils (1000/cubic mm)- Day140: number analyzed (Participants) | 2 | 10 | 0 | 0 | 0
  Neutrophils (1000/cubic mm)- Day140 | 2.01 [1.681 to 2.339] | 3.7175 [3.034 to 4.869] |  |  |
  Neutrophils (1000/cubic mm)- Day182: number analyzed (Participants) | 0 | 0 | 6 | 17 | 18
  Neutrophils (1000/cubic mm)- Day182 |  |  | 3.821 [3.278 to 4.284] | 3.264 [2.301 to 4.09] | 3.684 [2.86 to 4.14]
  Neutrophils (1000/cubic mm)- Day238: number analyzed (Participants) | 0 | 0 | 6 | 18 | 16
  Neutrophils (1000/cubic mm)- Day238 |  |  | 3.349 [2.832 to 3.886] | 3.413 [2.57 to 4.074] | 3.9935 [3.1115 to 4.3735]
  Neutrophils (1000/cubic mm)- Day334: number analyzed (Participants) | 0 | 0 | 6 | 18 | 16
  Neutrophils (1000/cubic mm)- Day334 |  |  | 3.3185 [2.85 to 3.559] | 3.135 [2.41 to 4.235] | 3.395 [2.7725 to 4.2395]

11. Primary Outcome: Number of Participants With Early Discontinuation of Vaccinations and Reason for Discontinuation
Description: From the study product discontinuation form, study product administration reasons are tabulated by treatment arm
Time Frame: Measured through study completion, up to 31 months
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Placebo | Part A: Vaccine | Part B: Placebo | Part B: Vaccine 1 | Part B: Vaccine 2
Number analyzed (Participants) | 2 | 10 | 6 | 21 | 21
Participants
  Adverse Experience | 0 | 0 | 0 | 0 | 1
  Reactogenicity Symptom | 0 | 0 | 0 | 1 | 0
  Unable to Contact/Out of Window | 0 | 0 | 0 | 0 | 5
  Participant Refused Vaccination | 0 | 0 | 0 | 1 | 1
  No Discontinuation | 2 | 10 | 6 | 19 | 14

12. Secondary Outcome: Occurrence of IgG HIV-1 Env-specific IgG Responses Two Weeks After the Last Vaccination
Description: Serum IgG responses were measured on a Bio-Plex instrument using a standardized custom Luminex assay. The readout is background-subtracted mean fluorescent intensity (MFI), with background adjustment for an antigen-specific plate level control. For each sample, response magnitude is net MFI, defined as experimental antigen MFI minus reference antigen MFI. Net MFI less than 1 is set to 1, and net MFI > 22,000 is set to 22,000. Samples from post-enrollment visits have positive responses if they meet three criteria: (1) net MFI greater than or equal to an antigen-specific response threshold (defined as the maximum of 100 and the 95th percentile of baseline net MFI), (2) net MFI values are greater than 3 times baseline net MFI, and (3) experimental antigen MFI values are greater than 3 times baseline MFI. Data are excluded if blood draw date was outside the allowable window, a participant was HIV-infected, reference antigen > 5,000 MFI, or baseline net MFI > 6,500.
Time Frame: Measured at Month 2.5 for part A and 8.5 for part B
Population: In this report, "Overall Number of Participants Analyzed" represents the HIV-uninfected participants who received the last vaccination with specimens at Month 2.5 for part A and Month 8.5 for part B. The "Number Analyzed" in the Outcome Measure Data Table shows the number of participants with available BAMA data after filtering for assay specific quality control criteria (excluding the reference antigen record which exceeds 5000 MFI etc.).
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Placebo | Part A: Vaccine | Part B: Placebo | Part B: Vaccine 1 | Part B: Vaccine 2
Number analyzed (Participants) | 2 | 10 | 6 | 19 | 16
Participants
  254008_D11gp120.avi/293F: number analyzed (Participants) | 2 | 8 | 6 | 19 | 15
  254008_D11gp120.avi/293F | 0 | 8 | 0 | 18 | 13
  51802_D11gp120.avi/293F: number analyzed (Participants) | 2 | 9 | 6 | 18 | 15
  51802_D11gp120.avi/293F | 0 | 9 | 0 | 18 | 13
  A244 D11gp120_avi: number analyzed (Participants) | 2 | 8 | 6 | 18 | 15
  A244 D11gp120_avi | 0 | 8 | 0 | 18 | 13
  B.6240_D11gp120/293F: number analyzed (Participants) | 2 | 9 | 6 | 19 | 15
  B.6240_D11gp120/293F | 0 | 9 | 0 | 17 | 13
  BJOX002_D11gp120.avi/293F: number analyzed (Participants) | 2 | 9 | 6 | 19 | 15
  BJOX002_D11gp120.avi/293F | 0 | 9 | 0 | 16 | 12
  BORI_D11gp120.avi/293F: number analyzed (Participants) | 2 | 10 | 6 | 19 | 15
  BORI_D11gp120.avi/293F | 0 | 9 | 0 | 15 | 11
  CNE20_D11gp120.avi/293F: number analyzed (Participants) | 2 | 8 | 6 | 18 | 15
  CNE20_D11gp120.avi/293F | 0 | 8 | 0 | 18 | 13
  TT31P.2792_D11gp120.avi/293F: number analyzed (Participants) | 2 | 8 | 6 | 18 | 15
  TT31P.2792_D11gp120.avi/293F | 0 | 8 | 0 | 18 | 13
  gp120-A: number analyzed (Participants) | 2 | 8 | 6 | 18 | 15
  gp120-A | 0 | 8 | 0 | 18 | 12
  gp120-AE: number analyzed (Participants) | 2 | 9 | 6 | 19 | 15
  gp120-AE | 0 | 9 | 0 | 17 | 13
  gp120-B: number analyzed (Participants) | 2 | 10 | 6 | 19 | 15
  gp120-B | 0 | 9 | 0 | 18 | 11
  gp120-C: number analyzed (Participants) | 2 | 9 | 6 | 19 | 15
  gp120-C | 0 | 9 | 0 | 17 | 12
  gp70-001428.2.42 V1V2: number analyzed (Participants) | 2 | 10 | 6 | 18 | 15
  gp70-001428.2.42 V1V2 | 0 | 6 | 0 | 17 | 11
  gp70-191084_B7 V1V2: number analyzed (Participants) | 2 | 9 | 6 | 18 | 15
  gp70-191084_B7 V1V2 | 0 | 9 | 0 | 17 | 11
  gp70-62357.14 V1V2: number analyzed (Participants) | 2 | 10 | 6 | 18 | 15
  gp70-62357.14 V1V2 | 0 | 5 | 0 | 14 | 9
  gp70-700010058 V1V2: number analyzed (Participants) | 2 | 10 | 6 | 18 | 15
  gp70-700010058 V1V2 | 0 | 1 | 0 | 15 | 11
  gp70-7060101641 V1V2: number analyzed (Participants) | 2 | 10 | 6 | 18 | 15
  gp70-7060101641 V1V2 | 0 | 6 | 0 | 17 | 10
  gp70-96ZM651.02 V1v2: number analyzed (Participants) | 2 | 10 | 6 | 18 | 15
  gp70-96ZM651.02 V1v2 | 0 | 8 | 0 | 16 | 11
  gp70-BF1266_431a_V1V2: number analyzed (Participants) | 2 | 10 | 6 | 18 | 15
  gp70-BF1266_431a_V1V2 | 0 | 5 | 0 | 17 | 8
  gp70-BJOX002000.03.2 V1V2: number analyzed (Participants) | 2 | 9 | 6 | 18 | 15
  gp70-BJOX002000.03.2 V1V2 | 0 | 8 | 0 | 17 | 11
  gp70-C2101.c01_V1V2: number analyzed (Participants) | 2 | 10 | 6 | 18 | 15
  gp70-C2101.c01_V1V2 | 0 | 6 | 0 | 17 | 11
  gp70-CAP210.2.00.E8 V1V2: number analyzed (Participants) | 2 | 10 | 6 | 18 | 15
  gp70-CAP210.2.00.E8 V1V2 | 0 | 6 | 0 | 16 | 8
  gp70-CM244.ec1 V1V2: number analyzed (Participants) | 2 | 8 | 6 | 18 | 15
  gp70-CM244.ec1 V1V2 | 0 | 8 | 0 | 18 | 11
  gp70-Ce1086_B2 V1V2: number analyzed (Participants) | 2 | 9 | 6 | 18 | 15
  gp70-Ce1086_B2 V1V2 | 0 | 8 | 0 | 18 | 13
  gp70-RHPA4259.7 V1V2: number analyzed (Participants) | 2 | 10 | 6 | 18 | 15
  gp70-RHPA4259.7 V1V2 | 0 | 5 | 0 | 16 | 8
  gp70-TT31P.2F10.2792 V1V2: number analyzed (Participants) | 2 | 10 | 6 | 18 | 15
  gp70-TT31P.2F10.2792 V1V2 | 0 | 4 | 0 | 13 | 9
  gp70-TV1.21 V1V2: number analyzed (Participants) | 2 | 10 | 6 | 18 | 15
  gp70-TV1.21 V1V2 | 0 | 7 | 0 | 17 | 9
  gp70_B.CaseA_V1_V2: number analyzed (Participants) | 2 | 10 | 6 | 18 | 15
  gp70_B.CaseA_V1_V2 | 0 | 6 | 0 | 17 | 11

13. Secondary Outcome: Levels of IgG HIV-1 Env-specific IgG Responses Two Weeks After the Last Vaccination
Description: Serum IgG responses were measured on a Bio-Plex instrument using a standardized custom Luminex assay. The readout is background-subtracted mean fluorescent intensity (MFI), with background adjustment for an antigen-specific plate level control. For each sample, response magnitude is net MFI, defined as experimental antigen MFI minus reference antigen MFI. Net MFI less than 1 is set to 1, and net MFI > 22,000 is set to 22,000. Data are excluded if blood draw date was outside the allowable window, a participant was HIV-infected, reference antigen > 5,000 MFI, or baseline net MFI > 6,500. Summary was calculated among positive responders only (positivity criteria are described in Outcome 12).
Time Frame: Measured at Month 2.5 for part A and 8.5 for part B
Population: as for outcome 12
Measure: Median (Inter-Quartile Range); unit: relative fluorescence units
Arm/Group | Part A: Vaccine | Part B: Vaccine 1 | Part B: Vaccine 2
Number analyzed (Participants) | 10 | 19 | 16
relative fluorescence units
  254008_D11gp120.avi/293F: number analyzed (Participants) | 8 | 18 | 13
  254008_D11gp120.avi/293F | 22000 [22000 to 22000] | 22000 [22000 to 22000] | 22000 [22000 to 22000]
  51802_D11gp120.avi/293F: number analyzed (Participants) | 9 | 18 | 13
  51802_D11gp120.avi/293F | 13847.8 [13546.5 to 22000] | 22000 [16922.6 to 22000] | 12427.5 [6267.8 to 22000]
  A244 D11gp120_avi: number analyzed (Participants) | 8 | 18 | 13
  A244 D11gp120_avi | 22000 [22000 to 22000] | 22000 [22000 to 22000] | 22000 [22000 to 22000]
  B.6240_D11gp120/293F: number analyzed (Participants) | 9 | 17 | 13
  B.6240_D11gp120/293F | 12265 [9028.5 to 18413.5] | 22000 [18193.8 to 22000] | 22000 [13876.8 to 22000]
  BJOX002_D11gp120.avi/293F: number analyzed (Participants) | 9 | 16 | 12
  BJOX002_D11gp120.avi/293F | 11645.2 [8450.2 to 15975.5] | 22000 [19076.4 to 22000] | 14547.1 [9620.1 to 21372.2]
  BORI_D11gp120.avi/293F: number analyzed (Participants) | 9 | 15 | 11
  BORI_D11gp120.avi/293F | 5944.5 [3552 to 8805.8] | 16031.8 [10413.1 to 20097] | 7429.2 [5766.5 to 12648.8]
  CNE20_D11gp120.avi/293F: number analyzed (Participants) | 8 | 18 | 13
  CNE20_D11gp120.avi/293F | 22000 [22000 to 22000] | 22000 [22000 to 22000] | 22000 [22000 to 22000]
  TT31P.2792_D11gp120.avi/293F: number analyzed (Participants) | 8 | 18 | 13
  TT31P.2792_D11gp120.avi/293F | 22000 [22000 to 22000] | 22000 [22000 to 22000] | 22000 [22000 to 22000]
  gp120-A: number analyzed (Participants) | 8 | 18 | 12
  gp120-A | 13589.6 [10025.8 to 18696.2] | 22000 [17859 to 22000] | 18287.8 [11116.1 to 21526.8]
  gp120-AE: number analyzed (Participants) | 9 | 17 | 13
  gp120-AE | 11629.5 [8498.8 to 13170.2] | 18609 [16413.8 to 22000] | 11534.5 [9247.5 to 19902.2]
  gp120-B: number analyzed (Participants) | 9 | 18 | 11
  gp120-B | 3895.2 [3754 to 8448.8] | 10957.1 [8435.3 to 16405.2] | 13483 [8970.9 to 19446.6]
  gp120-C: number analyzed (Participants) | 9 | 17 | 12
  gp120-C | 12084.8 [9242.8 to 17222] | 22000 [18300 to 22000] | 15846.6 [11677.2 to 22000]
  gp70-001428.2.42 V1V2: number analyzed (Participants) | 6 | 17 | 11
  gp70-001428.2.42 V1V2 | 4214.6 [1287.6 to 6912.2] | 3180 [1325.5 to 8855.8] | 7208.8 [3152.6 to 14312.9]
  gp70-191084_B7 V1V2: number analyzed (Participants) | 9 | 17 | 11
  gp70-191084_B7 V1V2 | 14985 [942 to 18635.2] | 21866.8 [13914.5 to 22000] | 21177.8 [10583.2 to 22000]
  gp70-62357.14 V1V2: number analyzed (Participants) | 5 | 14 | 9
  gp70-62357.14 V1V2 | 764.8 [247.8 to 3565.2] | 1399.8 [1077.1 to 3775.1] | 2140.8 [1302 to 3711.5]
  gp70-700010058 V1V2: number analyzed (Participants) | 1 | 15 | 11
  gp70-700010058 V1V2 | 3103 [3103 to 3103] | 2172.2 [396.2 to 6597.9] | 11938.2 [3265.8 to 22000]
  gp70-7060101641 V1V2: number analyzed (Participants) | 6 | 17 | 10
  gp70-7060101641 V1V2 | 402.6 [289.4 to 2538.8] | 1176.2 [842.5 to 2095.5] | 1217.4 [681.6 to 2033.7]
  gp70-96ZM651.02 V1v2: number analyzed (Participants) | 8 | 16 | 11
  gp70-96ZM651.02 V1v2 | 10010.6 [300.6 to 21457.8] | 12543.9 [8143.1 to 22000] | 11192.5 [6121.4 to 20222.1]
  gp70-BF1266_431a_V1V2: number analyzed (Participants) | 5 | 17 | 8
  gp70-BF1266_431a_V1V2 | 808 [560.2 to 5568.8] | 3456 [641 to 9020.8] | 2003.5 [1455.2 to 3187.4]
  gp70-BJOX002000.03.2 V1V2: number analyzed (Participants) | 8 | 17 | 11
  gp70-BJOX002000.03.2 V1V2 | 6452.2 [1076.9 to 11295.9] | 17549.8 [6772.8 to 22000] | 7962.2 [4547.6 to 15902.6]
  gp70-C2101.c01_V1V2: number analyzed (Participants) | 6 | 17 | 11
  gp70-C2101.c01_V1V2 | 14362 [5960.7 to 20792.3] | 11920.5 [6894 to 22000] | 7065.8 [2127.5 to 18989.5]
  gp70-CAP210.2.00.E8 V1V2: number analyzed (Participants) | 6 | 16 | 8
  gp70-CAP210.2.00.E8 V1V2 | 1596.2 [494.2 to 4094.9] | 1571.4 [487.8 to 5566.1] | 1641 [1030.9 to 2463.3]
  gp70-CM244.ec1 V1V2: number analyzed (Participants) | 8 | 18 | 11
  gp70-CM244.ec1 V1V2 | 22000 [18385.9 to 22000] | 22000 [22000 to 22000] | 22000 [13074.6 to 22000]
  gp70-Ce1086_B2 V1V2: number analyzed (Participants) | 8 | 18 | 13
  gp70-Ce1086_B2 V1V2 | 22000 [22000 to 22000] | 22000 [22000 to 22000] | 22000 [10914.2 to 22000]
  gp70-RHPA4259.7 V1V2: number analyzed (Participants) | 5 | 16 | 8
  gp70-RHPA4259.7 V1V2 | 782.5 [766.2 to 3177.2] | 2845.1 [1565.3 to 5682.8] | 1575.6 [1293.6 to 2538.4]
  gp70-TT31P.2F10.2792 V1V2: number analyzed (Participants) | 4 | 13 | 9
  gp70-TT31P.2F10.2792 V1V2 | 2308.4 [568.4 to 4841.8] | 1821.8 [1275.2 to 5421.5] | 1712.5 [1117.5 to 2679]
  gp70-TV1.21 V1V2: number analyzed (Participants) | 7 | 17 | 9
  gp70-TV1.21 V1V2 | 1249.8 [727.8 to 6326.6] | 3075.2 [636.5 to 8293.8] | 2528.5 [1957 to 3612.8]
  gp70_B.CaseA_V1_V2: number analyzed (Participants) | 6 | 17 | 11
  gp70_B.CaseA_V1_V2 | 1177 [613.9 to 5457.7] | 4071 [2531 to 10252.8] | 4955.8 [1717.6 to 13117.4]

14. Secondary Outcome: Breadth of IgG HIV-1 Env-specific IgG Responses Two Weeks After the Last Vaccination
Description: Serum IgG responses were measured on a Bio-Plex instrument using a standardized custom Luminex assay. Magnitude-breadth (MB) curves characterized the magnitude (Binding antibody MFI* at 1:50 dilution and titer) and breadth (number of antigens with positive response at given MFI* or titer) of each individual plasma sample assayed against a panel of antigens. The x-axis represents the response magnitude and the y-axis represents the fraction of antigens with response magnitude greater than the x-axis value. In addition to the individual sample specific curves, the group-specific curve displayed the average MB across all participants in that group. The area-under-the-magnitude-breadth curve (AUC-MB) was calculated as the average of the log10 MFI* (log10 titer) over the panel of antigens.
Time Frame: Measured at Month 2.5 for part A and 8.5 for part B
Population: as for outcome 12
Measure: Median (Inter-Quartile Range); unit: log10 titer* proportion of antigens
Arm/Group | Part A: Placebo | Part A: Vaccine | Part B: Placebo | Part B: Vaccine 1 | Part B: Vaccine 2
Number analyzed (Participants) | 2 | 10 | 6 | 19 | 16
log10 titer* proportion of antigens
  gp120 Breadth Panel: number analyzed (Participants) | 2 | 8 | 6 | 18 | 15
  gp120 Breadth Panel | 2 [2 to 2] | 4 [3.9 to 4.1] | 2 [2 to 2] | 4.2 [4.1 to 4.4] | 4 [3.4 to 4.1]
  gp70 V1V2 Breadth Panel: number analyzed (Participants) | 2 | 8 | 6 | 18 | 15
  gp70 V1V2 Breadth Panel | 2 [2 to 2] | 2.7 [2.5 to 3.1] | 2 [2 to 2] | 3.3 [3 to 3.6] | 3.2 [2.3 to 3.5]

15. Secondary Outcome: Part B: Occurrence of Serum Neutralizing Antibody Responses Against Tier 1A, Tier 1B, and Selected Tier 2 Viruses Two Weeks After the Last Vaccination
Description: Neutralizing antibodies against HIV1were measured as a function of reductions in Tat-regulatedluciferase (Luc) reporter gene expression in TZM-blcells. The assay performed in TZM-bl cells measured neutralization titers against a panel of Env-pseudotyped viruses that exhibit the following naturalization phenotypes. Response to a virus/isolate was considered positive if the neutralization titer was above a prespecified cutoff. A titer was defined as the serum dilution that reduced relative luminescence units (RLUs) by 50% and 80% relative to the RLUs in virus control wells (cells + virus only) after subtraction of background RLU (ID50 and ID80, cells only). The prespecified cutoff was 20 for MW965.26 (Tier 1a) and 10 for other viruses.
Time Frame: Measured at Month 8.5 for part B only
Population: In this report, "Overall Number of Participants Analyzed" represents the HIV-uninfected participants who received the last vaccination with specimens at Month 2.5 for part A and Month 8.5 for part B. The "Number Analyzed" in the Outcome Measure Data Table shows the number of participants with available Neutralizing Antibody data after filtering for assay specific quality control criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: Placebo | Part B: Vaccine 1 | Part B: Vaccine 2
Number analyzed (Participants) | 6 | 19 | 16
Participants
  MW965.26 (ID50) | 0 | 16 | 15
  1056-10.TA11.1826 (ID50) | 0 | 0 | 0
  6535.3 (ID50) | 0 | 0 | 0
  Bx08.16 (ID50) | 0 | 3 | 0
  Q23.17 (ID50) | 0 | 0 | 0
  ZM197M.PB7 (ID50) | 0 | 0 | 0
  92UG037.1 (ID50) | 0 | 0 | 2
  JR-FL (ID50) | 0 | 0 | 0
  MW965.26 (ID80) | 0 | 16 | 14
  1056-10.TA11.1826 (ID80) | 0 | 0 | 0
  6535.3 (ID80) | 0 | 0 | 0
  Bx08.16 (ID80) | 0 | 0 | 0
  Q23.17 (ID80) | 0 | 0 | 0
  ZM197M.PB7 (ID80) | 0 | 0 | 0
  92UG037.1 (ID80) | 0 | 0 | 0
  JR-FL (ID80) | 0 | 0 | 0

16. Secondary Outcome: Part B: Levels of Serum Neutralizing Antibody Responses Against Tier 1A, Tier 1B, and Selected Tier 2 Viruses Two Weeks After the Last Vaccination
Description: as for outcome 15
Time Frame: Measured at Month 8.5 for part B only
Population: as for outcome 15
Measure: Median (Inter-Quartile Range); unit: Titers
Arm/Group | Part B: Placebo | Part B: Vaccine 1 | Part B: Vaccine 2
Number analyzed (Participants) | 6 | 19 | 16
Titers
  MW965.26 (ID50) | 10 [10 to 10] | 681.2 [327.4 to 906.1] | 583.5 [227.2 to 1306.6]
  1056-10.TA11.1826 (ID50) | 5 [5 to 5] | 5 [5 to 5] | 5 [5 to 5]
  6535.3 (ID50) | 5 [5 to 5] | 5 [5 to 5] | 5 [5 to 5]
  Bx08.16 (ID50) | 5 [5 to 5] | 5 [5 to 5] | 5 [5 to 5]
  Q23.17 (ID50) | 5 [5 to 5] | 5 [5 to 5] | 5 [5 to 5]
  ZM197M.PB7 (ID50) | 5 [5 to 5] | 5 [5 to 5] | 5 [5 to 5]
  92UG037.1 (ID50) | 5 [5 to 5] | 5 [5 to 5] | 5 [5 to 5]
  JR-FL (ID50) | 5 [5 to 5] | 5 [5 to 5] | 5 [5 to 5]
  MW965.26 (ID80) | 10 [10 to 10] | 233.7 [100.9 to 331] | 181 [74.2 to 426.3]
  1056-10.TA11.1826 (ID80) | 5 [5 to 5] | 5 [5 to 5] | 5 [5 to 5]
  6535.3 (ID80) | 5 [5 to 5] | 5 [5 to 5] | 5 [5 to 5]
  Bx08.16 (ID80) | 5 [5 to 5] | 5 [5 to 5] | 5 [5 to 5]
  Q23.17 (ID80) | 5 [5 to 5] | 5 [5 to 5] | 5 [5 to 5]
  ZM197M.PB7 (ID80) | 5 [5 to 5] | 5 [5 to 5] | 5 [5 to 5]
  92UG037.1 (ID80) | 5 [5 to 5] | 5 [5 to 5] | 5 [5 to 5]
  JR-FL (ID80) | 5 [5 to 5] | 5 [5 to 5] | 5 [5 to 5]

17. Secondary Outcome: Breadth of gp70-V1V2 IgG and gp120 IgA, Assessed by Binding Antibody Multiplex Assay, and ADCC Activities Against HIV-1 Subtypes A, B, C and A/E Two Weeks After the Last Vaccination in Part B
Description: For Binding Antibody Multiplex Assay, gp70-V1V2 IgG, the area-under-the-magnitude-breadth curve (AUC-MB) was calculated as the average of the log10 MFI* (log10 titer) over the panel of antigens. For ADCC GranToxiLux, AUC-MB was calculated as the average of the AUC over the panel of antigens, where AUC is defined as nonparametric area under the net percent granzyme B activity vs log10 (dilution) curve ("AUC"), calculated using the trapezoidal rule, and setting any net percent granzyme B activity below 0% to 0%. For ADCC Luciferase, (AUC-MB) was calculated as the average of the pAUC over the panel of antigens, where pAUC is defined as nonparametric partial area under the baseline subtracted curves ("pAUC"), calculated using the trapezoidal rule on the first four dilutions of the baseline subtracted curves, setting baseline subtracted loss Luciferase activity less than 0% to zero.
Time Frame: Measured at Month 8.5 for part B only
Population: In this report, "Overall Number of Participants Analyzed" represents the HIV-uninfected participants who received the last vaccination with specimens at Month 8.5 for part B. The "Number Analyzed" in the Outcome Measure Data Table shows the number of participants with available BAMA, or ADCC data after filtering for assay specific quality control criteria. Assay data were not collected for gp120 IgA per lab study plan.
Measure: Median (Inter-Quartile Range); unit: log10 titer* proportion of antigens
Arm/Group | Part B: Placebo | Part B: Vaccine 1 | Part B: Vaccine 2
Number analyzed (Participants) | 6 | 19 | 16
log10 titer* proportion of antigens
  ADCC GranToxiLux against HIV-1 subtypes A, B, C and A/E | 0.2 [0.1 to 0.6] | 19 [13.9 to 25] | 11.4 [7.1 to 16.3]
  ADCC Luciferase against HIV-1 subtypes A, B, C and A/E | 2.2 [1.3 to 2.9] | 31.8 [19.3 to 45.8] | 17.8 [10.5 to 28.7]
  gp70 V1V2 IgG: number analyzed (Participants) | 6 | 18 | 15
  gp70 V1V2 IgG | 2 [2 to 2] | 3.3 [3 to 3.6] | 3.2 [2.3 to 3.5]
  gp120 IgA: number analyzed (Participants) | 0 | 0 | 0

18. Secondary Outcome: Occurrence of CD4+ T Cell Responses to the HIV Proteins Included in the Vaccine Two Weeks After the Last Vaccination. Measured by Flow Cytometry.
Description: PBMC samples are stimulated with synthetic peptide pools or left unstimulated as a negative control. For each sample, T-cell subset, and peptide pool, response magnitude is % cells expressing markers (IFNg and/or IL-2) after peptide stimulation minus % cells expressing markers after no stimulation. A contingency table is constructed to assess response: stimulation (peptide/none) vs. marker expression (yes/no). A one-sided Fisher's exact test is applied, testing if the number of cells positive for the marker is equal in the stimulated vs. unstimulated cells. A discrete Bonferroni adjustment is made over the peptide pools. Response is positive if adjusted p-value <=0.00001. Please note the above analyses were applied by the lab to determine the response positivity, not the planned analyses for the study outcome measures. Data are excluded if blood draw date was outside the visit window, participant was HIV-infected, PBMC viability or T-cell count were low, or negative control was high.
Time Frame: Measured at Month 8.5 for part B only
Population: In this report, "Overall Number of Participants Analyzed" represents the HIV-uninfected participants who received the last vaccination with specimens at Month 8.5 for part B. The "Number Analyzed" in the Outcome Measure Data Table shows the number of participants with available ICS data after filtering for assay specific quality control criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: Placebo | Part B: Vaccine 1 | Part B: Vaccine 2
Number analyzed (Participants) | 6 | 19 | 16
Participants
  ANY ENV PTEG | 0 | 19 | 7
  ANY GAG PTEG | 0 | 1 | 0
  ENV-1-PTEG-SEQ | 0 | 17 | 7
  ENV-2-PTEG-SEQ | 0 | 16 | 4
  GAG-1-PTEG-SEQ | 0 | 0 | 0
  GAG-2-PTEG-SEQ | 0 | 1 | 0

19. Secondary Outcome: Level of CD4+ T Cell Responses to the HIV Proteins Included in the Vaccine Two Weeks After the Last Vaccination. Measured by Flow Cytometry.
Description: as for outcome 18
Time Frame: Measured at Month 8.5 for part B only
Population: as for outcome 18
Measure: Median (Inter-Quartile Range); unit: % CD4+ T-cells
Arm/Group | Part B: Placebo | Part B: Vaccine 1 | Part B: Vaccine 2
Number analyzed (Participants) | 6 | 19 | 16
% CD4+ T-cells
  ANY ENV PTEG | -0.011 [-0.015 to -0.008] | 0.313 [0.183 to 0.386] | 0.102 [0.053 to 0.236]
  ANY GAG PTEG | -0.001 [-0.007 to 0.003] | 0.017 [-0.004 to 0.028] | 0.001 [-0.006 to 0.009]
  ENV-1-PTEG-SEQ | -0.005 [-0.009 to -0.003] | 0.166 [0.1 to 0.209] | 0.052 [0.026 to 0.131]
  ENV-2-PTEG-SEQ | -0.007 [-0.01 to -0.004] | 0.142 [0.064 to 0.194] | 0.037 [0.019 to 0.058]
  GAG-1-PTEG-SEQ | -0.001 [-0.003 to 0.003] | 0.004 [-0.004 to 0.018] | -0.002 [-0.008 to 0.005]
  GAG-2-PTEG-SEQ | -0.002 [-0.004 to 0.001] | 0.009 [0 to 0.017] | 0.003 [-0.002 to 0.006]

20. Secondary Outcome: Occurrence of CD8+ T Cell Responses to the HIV Proteins Included in the Vaccine Two Weeks After the Last Vaccination. Measured by Flow Cytometry.
Description: as for outcome 18
Time Frame: Measured at Month 8.5 for part B only
Population: as for outcome 18
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: Placebo | Part B: Vaccine 1 | Part B: Vaccine 2
Number analyzed (Participants) | 6 | 19 | 16
Participants
  ANY ENV PTEG: number analyzed (Participants) | 5 | 19 | 16
  ANY ENV PTEG | 0 | 0 | 0
  ANY GAG PTEG: number analyzed (Participants) | 5 | 19 | 16
  ANY GAG PTEG | 0 | 0 | 0
  ENV-1-PTEG-SEQ: number analyzed (Participants) | 5 | 19 | 16
  ENV-1-PTEG-SEQ | 0 | 0 | 0
  ENV-2-PTEG-SEQ: number analyzed (Participants) | 5 | 19 | 16
  ENV-2-PTEG-SEQ | 0 | 0 | 0
  GAG-1-PTEG-SEQ: number analyzed (Participants) | 5 | 19 | 16
  GAG-1-PTEG-SEQ | 0 | 0 | 0
  GAG-2-PTEG-SEQ: number analyzed (Participants) | 5 | 19 | 16
  GAG-2-PTEG-SEQ | 0 | 0 | 0

21. Secondary Outcome: Level of CD8+ T Cell Responses to the HIV Proteins Included in the Vaccine Two Weeks After the Last Vaccination. Measured by Flow Cytometry.
Description: as for outcome 18
Time Frame: Measured at Month 8.5 for part B only
Population: as for outcome 18
Measure: Median (Inter-Quartile Range); unit: % CD8+ T-cells
Arm/Group | Part B: Placebo | Part B: Vaccine 1 | Part B: Vaccine 2
Number analyzed (Participants) | 6 | 19 | 16
% CD8+ T-cells
  ANY ENV PTEG: number analyzed (Participants) | 5 | 19 | 16
  ANY ENV PTEG | -0.003 [-0.008 to 0.004] | 0.007 [-0.002 to 0.013] | -0.007 [-0.012 to 0]
  ANY GAG PTEG: number analyzed (Participants) | 5 | 19 | 16
  ANY GAG PTEG | 0.002 [-0.011 to 0.003] | -0.006 [-0.009 to 0.002] | -0.004 [-0.013 to -0.001]
  ENV-1-PTEG-SEQ: number analyzed (Participants) | 5 | 19 | 16
  ENV-1-PTEG-SEQ | 0.001 [-0.003 to 0.004] | 0.006 [-0.001 to 0.017] | -0.002 [-0.007 to 0.002]
  ENV-2-PTEG-SEQ: number analyzed (Participants) | 5 | 19 | 16
  ENV-2-PTEG-SEQ | -0.002 [-0.007 to 0] | 0 [-0.008 to 0.007] | -0.004 [-0.006 to 0]
  GAG-1-PTEG-SEQ: number analyzed (Participants) | 5 | 19 | 16
  GAG-1-PTEG-SEQ | 0.002 [-0.009 to 0.007] | 0 [-0.004 to 0.002] | -0.005 [-0.009 to 0]
  GAG-2-PTEG-SEQ: number analyzed (Participants) | 5 | 19 | 16
  GAG-2-PTEG-SEQ | 0 [-0.003 to 0.001] | -0.004 [-0.007 to 0] | 0 [-0.005 to 0.002]

ADVERSE EVENTS:
Time Frame: Serious Adverse events are collected throughout the study (months 0-8 for Part A, and months 0-14 for Part B). Non-serious adverse events are collected through 30 days after each vaccination (at months 0,2 for Part A, and months 0, 1, 3, 6, 8 for Part B).
Arm/Group | Part A: Placebo | Part A: Vaccine | Part B: Placebo | Part B: Vaccine 1 | Part B: Vaccine 2
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/10 | 0/6 | 0/21 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/10 | 0/6 | 0/21 | 0/21
Other Adverse Events (participants affected / at risk) | 2/2 | 6/10 | 5/6 | 19/21 | 18/21
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: Placebo (N=2) | Part A: Vaccine (N=10) | Part B: Placebo (N=6) | Part B: Vaccine 1 (N=21) | Part B: Vaccine 2 (N=21)
Any Event in SOC (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Lymph node pain (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Any Event in SOC (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eustachian tube dysfunction (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Any Event in SOC (Gastrointestinal disorders) | 0 (0) | 1 (1) | 4 (4) | 5 (5) | 3 (5)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anal fissure (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anal fissure haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cannabinoid hyperemesis syndrome (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 2 (2)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tongue ulceration (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Any Event in SOC (General disorders) | 0 (0) | 0 (0) | 1 (1) | 4 (5) | 1 (2)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cyst (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injection site pruritus (General disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (2)
Any Event in SOC (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatic cyst (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Any Event in SOC (Infections and infestations) | 0 (0) | 3 (3) | 3 (4) | 10 (18) | 13 (25)
Abscess limb (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Body tinea (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchitis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Febrile infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Otitis media (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tooth abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2) | 1 (2) | 8 (9) | 10 (13)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Vulvovaginal mycotic infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Any Event in SOC (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1) | 3 (4) | 0 (0)
Chest injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Nasal injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Post procedural swelling (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Any Event in SOC (Investigations) | 0 (0) | 3 (4) | 1 (1) | 5 (8) | 4 (6)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 2 (2) | 1 (1) | 4 (4) | 4 (4)
Blood glucose increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Red blood cells urine positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Any Event in SOC (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 5 (5) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Any Event in SOC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemangioma of liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Any Event in SOC (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Tardive dyskinesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Any Event in SOC (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nightmare (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Panic attack (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Any Event in SOC (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (2) | 2 (2) | 2 (4)
Glycosuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 2 (3)
Any Event in SOC (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Menorrhagia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Any Event in SOC (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Any Event in SOC (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (2) | 1 (1) | 4 (5) | 5 (6)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Papule (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Any Event in SOC (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-09-28): https://cdn.clinicaltrials.gov/large-docs/76/NCT03409276/Prot_000.pdf
  • Statistical Analysis Plan (2021-01-25): https://cdn.clinicaltrials.gov/large-docs/76/NCT03409276/SAP_001.pdf